CLINICAL TRIAL: NCT00151710
Title: Effects of Pioglitazone in Glucocorticoid-Induced Insulin Resistance. Studies in Congenital Adrenal Hyperplasia.
Brief Title: Effects of Pioglitazone in Congenital Adrenal Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H6E-UT-O013
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
Congenital adrenal hyperplasia, an autosomal recessive condition, is mainly caused by mutations in the gene 21-hydroxylase and is treated with glucocorticoids in a slightly supraphysiological dose. Adult patients seem to be characterized by insulin resistance, which may be caused by the glucocorticoids and/or the accompanying obesity. The hypothesis of this study is that pioglitazone can improve insulin sensitivity and correlated cardiovascular risk factors in this specific group of patients. This will be tested in a randomized, placebo-controlled, cross-over trial; insulin sensitivity will be quantified by euglycemic hyperinsulinemic clamp studies.

ELIGIBILITY:
Inclusion Criteria:

* biochemical and genetically proven congenital adrenal hyperplasia
* stable corticosteroid replacement for 3 months

Exclusion Criteria:

* age < 18 years
* inability to give informed consent
* significant cardiovascular disease, defined as myocardial infarction or stroke, six months preceding the study
* significant renal disease, GFR < 30 ml/min
* significant liver disease, defined as more than 3 times upper limit of normal values of alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
* pregnancy
* mental disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis J Tack, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands